CLINICAL TRIAL: NCT02428985
Title: Drug Use Investigation of Riociguat for Pulmonary Arterial Hypertension (PAH)
Brief Title: Prospective, Non-interventional, Multi-center, Post-authorization Safety Study of Riociguat for Pulmonary Arterial Hypertension (PAH)
Acronym: JPMS-PAH
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 17519; AD1510JP (Other: Company Internal)
Record Dates: First submitted 2015-04-21; First posted 2015-04-29 (Estimated); Last update posted 2024-01-29 (Actual); Status verified 2024-01

CONDITIONS: Hypertension, Pulmonary
Keywords: Riociguat; Adempas; soluble guanylate cyclase (sGC) stimulator; Pulmonary arterial hypertension; Japan; Post-marketing surveillance
MeSH Terms: conditions — Hypertension, Pulmonary; Limb-girdle muscular dystrophy, type 2E; Pulmonary Arterial Hypertension | interventions — riociguat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Riociguat: Riociguat treatment group
  Interventions: Drug: Riociguat (ADEMPAS, BAY63-2521)

INTERVENTIONS:
Drug: Riociguat (ADEMPAS, BAY63-2521) — The treatment of Riociguat should comply with the local product information

SUMMARY:
The primary objective in this study is to collect post-marketing information on Riociguat safety.Thus, the information on adverse events (AEs) and adverse drug reactions (ADRs) that occur within the first 12 months and in the following 6 -year observation at most, after starting Riociguat treatment under the routine clinical practice will be collected.

The secondary objectives are collecting information on Riociguat effectiveness, such as 6-Minute Walking Distance (6MWD) Test. Since it is assumed that Riociguat is for long-term use, information on Pulmonary Arterial Hypertension (PAH) clinical worsening will also be surveyed once a year.

DETAILED DESCRIPTION:
This local, prospective, non-interventional, multi-center study includes patients treated with Riociguat for PAH. A total of 600 patients (valid for safety analysis) is planned to be included in 4 years. This study is performed as an "all-case investigation" therefore; all patients who receive Riociguat treatment for PAH need to be registered, in principle. The treatment should be performed based on the product label in Japan. The standard observation period will last for 12 months from starting Riociguat treatment. Safety and effectiveness will be evaluated at the 3rd and 12th month of treatment. In addition, the extension observation period will be carried out as long as Riociguat treatment continues or at most for more 6 years. The purpose is to collect information on safety and effectiveness, such as adverse events and clinical worsening of PAH, once a year. Combining the standard observation and the extension observation period the patient could be followed for at most 7 years. When Riociguat treatment is terminated, the observation of the patient ends. The investigator should record data for each patient, as defined in the protocol, using the Electronic Data Capture (EDC) system. The duration of the study is of approximately 8 years from PAH indication approval.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are treated with Riociguat for PAH

Exclusion Criteria:

* N/A

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population includes patients treated with Riociguat for PAH. This study is performed as an all-case investigation. Therefore, all patients who have been treated with Riociguat for PAH need to be registered in principle, until the target number of patients reached.
Sampling Method: Non-Probability Sample
Enrollment: 882 (Actual)
Dates: Start 2015-06-29 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment emergent adverse events. Adverse events of special interest:Hypotension,Gastrointestinal disorder,Hemoptysis, pulmonary hemorrhage and Pulmonary congestion, pulmonary edema | Up to 7 years
Number of participants with adverse drug reaction | Up to 7 years

SECONDARY OUTCOMES:
Change from baseline in 6-Minute Walking Distance at 3 months and 12 months | Baseline and 3 months,Baseline and 12 months
Change from baseline in Pulmonary Vascular Resistance (PVR) after 3 and 12 months | Baseline and 3 months,Baseline and 12 months
Change from baseline in tricuspid regurgitation pressure gradient (TRPG) after 3 and 12 months | Baseline and 3 months,Baseline and 12 months
Change in blood concentration from baseline in brain natriuretic peptide / N-terminal pro-brain natriuretic peptide (BPN/NT-pro BNP) after 3 and 12 months. | Baseline and 3 months,Baseline and 12 months
Change from baseline in WHO functional class after 3 and 12 months | Baseline and 3 months,Baseline and 12 months
Time to Clinical Worsening | Up to 7 years
  The 1st occurrence of the following events is recorded & will considered for the calculation of the combined endpoint : -Death (all-cause mortality)-Heart/lung transplantation -Atrial Septostomy -Hospitalization due to persistent worsening of Pulmonary Hypertension -Start of new PH specific treatment (endothelin receptor antagonists, prostacycline analogues)or modification of a preexisting Prostacycline analogues treatment)due to worsening Pulmonary Hypertension (WPH) -Persistent decrease in 6MWD due to WPH (e.g. more than 15 % from baseline or more than 30% compared to the last measurement)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Multiple Locations, Japan

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.